CLINICAL TRIAL: NCT01448317
Title: A Randomized, Double-Blind, Placebo-Controlled, Ascending Single-Dose Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Subcutaneously Administered SAR236553 in Japanese Healthy Male Subjects
Brief Title: Ascending Dose Study of the Safety and Tolerability of Alirocumab (SAR236553/REGN727) in Japanese Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TDU12190; U1111-1118-1213 (Other: UTN)
Record Dates: First submitted 2011-09-21; First posted 2011-10-07 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — alirocumab; Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Experimental): Alirocumab dose 1 versus placebo
  Interventions: Drug: Alirocumab (Lyophilized formulation); Drug: Placebo (Lyophilized formulation)
- Cohort 2 (Experimental): Alirocumab dose 2 versus placebo
  Interventions: Drug: Alirocumab (Lyophilized formulation); Drug: Placebo (Lyophilized formulation)
- Cohort 3 (Experimental): Alirocumab dose 3 versus placebo
  Interventions: Drug: Alirocumab (Lyophilized formulation); Drug: Placebo (Lyophilized formulation)
- Cohort 4 (Experimental): Alirocumab dose 4 versus placebo
  Interventions: Drug: Alirocumab (Solution); Drug: Placebo (Solution)

INTERVENTIONS:
Drug: Alirocumab (Solution) — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Other Names: SAR236553; REGN727
  Arms: Cohort 4
Drug: Alirocumab (Lyophilized formulation) — Pharmaceutical form: lyophilized formulation
  Route of administration: subcutaneous
  Other Names: SAR236553; REGN727
  Arms: Cohort 1; Cohort 2; Cohort 3
Drug: Placebo (Solution) — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Arms: Cohort 4
Drug: Placebo (Lyophilized formulation) — Pharmaceutical form: lyophilized formulation
  Route of administration: Subcutaneous
  Arms: Cohort 1; Cohort 2; Cohort 3

SUMMARY:
Primary Objective:

To assess the safety and tolerability of ascending single doses of subcutaneously (SC) administered alirocumab (SAR236553/REGN727) in Japanese healthy male subjects.

Secondary Objectives:

* To assess the pharmacodynamics effect of a single SC dose of alirocumab on serum low-density lipoprotein cholesterol (LDL-C) and other lipids and apolipoproteins such as total cholesterol, high-density lipoprotein cholesterol (HDL-C), non-high-density lipoprotein cholesterol, very low-density lipoprotein cholesterol, Triglycerides, Apolipoprotein B, Apolipoprotein A1 and Lipoprotein(a).
* To assess the Pharmacokinetic profile of a single SC dose of alirocumab.
* To assess the immunogenicity of a single SC dose of alirocumab.

DETAILED DESCRIPTION:
4 sequential dose cohorts. Single dose followed by a total observation period of 15 weeks (106 days) for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subject, between 20 and 65 years inclusive.
* Body weight between 50.0 and 95.0 kg inclusive, body mass index between 18.0 and 30.0 kg/m² inclusive.
* Serum LDL-C levels >100 mg/dL

Exclusion Criteria:

* Subject indicated for the use of statins according to criteria in Adult Treatment Panel (ATP) III Guidelines as updated in 2004
* Significant concomitant illness or history of significant illness such as cardiac, renal, neurological, endocrinological, dermatological, metabolic or lymphatic disease, or any other illness or condition that would adversely affect the subject's participation in this study.
* History or presence of drug or alcohol abuse
* Smoking more than 5 cigarettes or equivalent in any 24 hour period.
* Any medication (including St John's Wort) within 14 days before the inclusion or within 5 times the elimination half-life or pharmacodynamic (PD) half-life of that drug, whichever the longest; any vaccination within the last 28 days.
* Positive reaction to any of the following tests: hepatitis B surface (HBs Ag) antigen, anti-hepatitis B core antibodies (anti-HBc Ab), anti-hepatitis C virus (anti-HCV) antibodies, human immunodeficiency virus (HIV) antigen and antibodies, syphilis.
* Elevated cholesterol due to a secondary cause such as hypothyroidism or alcohol.
* Presence or history of drug hypersensitivity
* Initiation of a new exercise routine or major change to a previous exercise routine within 4 weeks prior to Screening.
* Initiation of a new diet or major change to a previous diet within 4 weeks prior to Screening.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-05; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events | 106 days

SECONDARY OUTCOMES:
Change in serum Low-Density Lipoprotein Cholesterol (LDL-C) from baseline to each visit. | 106 days
Change in ApolipoproteinB, ApolipoproteinA1 and Lipoprotein(a) from baseline to each visit. | 106 days
Change in Total Cholesterol (T-C), High-Density Lipoprotein Cholesterol (HDL-C), Very Low-Density Lipoprotein Cholesterol (VLDL-C) and Triglycerides (TG) from baseline to each visit. | 106 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Tokyo, Japan

REFERENCES:
- [Result] Teramoto T, Kobayashi M, Uno K, Takagi Y, Matsuoka O, Sugimoto M, Inoue S, Minami F, Baccara-Dinet MT. Efficacy and Safety of Alirocumab in Japanese Subjects (Phase 1 and 2 Studies). Am J Cardiol. 2016 Jul 1;118(1):56-63. doi: 10.1016/j.amjcard.2016.04.011. Epub 2016 Apr 21. PMID 27184170